CLINICAL TRIAL: NCT06283017
Title: Acute Proof-of-Concept Study to Evaluate Hypoglossal Nerve Stimulation in Humans With Obstructive Sleep Apnea
Brief Title: Evaluation of the Effects of Hypoglossal Nerve Stimulation in Humans With Obstructive Sleep Apnea
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Invicta Medical Inc. (Industry)
Collaborators: Adelaide Institute for Sleep Health, Flinders University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IM-002
Record Dates: First submitted 2024-02-13; First posted 2024-02-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Sleep Apnea; Sleep Apnea, Obstructive; Sleep Disorder; Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hypoglossal nerve stimulation (Experimental): Device-mediated stimulation of the hypoglossal nerve
  Interventions: Device: Hypoglossal nerve stimulation

INTERVENTIONS:
Device: Hypoglossal nerve stimulation — Device stimulation of the hypoglossal nerve

SUMMARY:
This proof-of-concept study is being performed to evaluate whether the hypoglossal nerve can be stimulated using a small series of electrodes placed surgically via a percutaneous approach. Minimally invasive off the shelf medical devices will be used and observation of the characteristic physiological responses to stimulation of the HGN, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Subject must be eligible for a diagnostic or surgical procedure and

* Suffers from OSA (apnea/hypopnea index >10 event/h sleep) based on history and a physical exam.
* Is a surgical candidate.
* Is willing and capable of providing informed consent.
* Is willing to have a representative electrode array temporarily placed in the submandibular and mylohyoid space.
* Is willing to participate in the designated follow-up visits.
* Must be in good general health.
* Is able to understand and has voluntarily signed and dated the IRB or EC approved informed consent form (ICF) prior to initiation of any screening or study-specific procedure.
* Must be minimum of 18 years and maximum 80 years of age.

Exclusion Criteria:

* Has Body Mass Index above 35 kg/m2.
* Has had surgical resection or radiation therapy for cancer or congenital malformations in the larynx, tongue, or throat.
* Has significant co-morbidities making them unable or inappropriate to participate in this POC study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Target identification and access outcomes | Day 0
  Identification of and access to the target stimulation location aligned with the medial branch of the Hypoglossal Nerve
Tongue protrusion outcomes | Day 0
  Visual verification of protrusion of the tongue during stimulation at the target stimulation location with a representative electrode array.
Characterization of lead placement outcomes | Day 0
  Spatial characterization of the orientation of the electrode array and lead body to the target stimulation location considering suitable chronic anchoring locations.
Lead placement and removal outcomes | Day 0
  To demonstrate the ability to safely place and remove the electrode array, per protocol instructions.
Safety outcomes | Day 30
  To evaluate and report all observed adverse events, serious adverse events, unanticipated adverse events and adverse device effects observed during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Adelaide Institute for Sleep Health, Flinders University, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No